CLINICAL TRIAL: NCT05766514
Title: Phase II Prospective Randomized Control Trial of Cladribine and Low-Dose Cytarabine (LoDAC) Alternating With Decitabine vs. Hypomethylating Agents (HMA) Plus Venetoclax as Frontline Therapy for AML or High-Grade MDS in Patients Unfit for Intensive Induction
Brief Title: Trial of Cladribine and Low-Dose Cytarabine (LoDAC) Alternating With Decitabine vs. Hypomethylating Agents (HMA) Plus Venetoclax as Frontline Therapy for AML or High-Grade MDS in Patients Unfit for Intensive Induction
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study disapproved by internal scientific review committee on re-review; study will no longer move forward
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF-HEM-011; OCR43074 (Other: University of Florida); IRB202300983 (Other: University of Florida)
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: acute myeloid leukemia; myelodysplastic syndrome; AML; MDS; induction therapy; low-dose cytarabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Cladribine; Cytarabine; Decitabine; Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (investigational arm): cladribine, cytarabine, and decitabine (Experimental)
  Interventions: Drug: Cladribine; Drug: Cytarabine; Drug: Decitabine
- Arm B (control arm): azacitidine with venetoclax or decitabine with venetoclax (Active Comparator)
  Interventions: Drug: azacitidine or decitabine; Drug: Venetoclax

INTERVENTIONS:
Drug: Cladribine — Subjects will be given 5 mg/m2 cladribine intravenously on days 1-5 of cycle 1 and on days 1-3 of cycles 2, 5, 6, 9, 10, 13, 14, 17 and 18.
  Arms: Arm A (investigational arm): cladribine, cytarabine, and decitabine
Drug: Cytarabine — Subjects will be given 20 mg cytarabine subcutaneously twice daily on days 1-10 of cycles 1, 2, 5, 6, 9, 10, 13, 14, 17 and 18.
  Arms: Arm A (investigational arm): cladribine, cytarabine, and decitabine
Drug: Decitabine — Subjects will be given 20 mg/m2 decitabine intravenously on days 1-5 of cycles 3, 4, 7, 8, 11, 12, 15 and 16
  Arms: Arm A (investigational arm): cladribine, cytarabine, and decitabine
Drug: azacitidine or decitabine — Subjects will be given either 20 mg/m2 decitabine intravenously on days 1-5 of each cycle or 75 mg/m2 azacitidine intravenously or subcutaneously on days 1-7 of each cycle. The treating physician will determine which drug each subject will receive.
  Arms: Arm B (control arm): azacitidine with venetoclax or decitabine with venetoclax
Drug: Venetoclax — Subject will take 400 mg venetoclax orally once daily on days 1-21 of each cycle.
  Arms: Arm B (control arm): azacitidine with venetoclax or decitabine with venetoclax

SUMMARY:
This phase II, open-label, randomized trial will compare the efficacy of the novel regimen of cladribine/low-dose cytarabine alternating with decitabine to the current standard of care regimen of hypomethylating agents (decitabine or azacitidine) plus venetoclax in patients with acute myeloid leukemia (AML) or high-grade myelodysplastic syndrome (MDS) who are either elderly or unfit for intensive induction. Subjects will be randomized to be treated with either cladribine/low-dose cytarabine alternating with decitabine (Arm A) or decitabine or azacitadine plus venetoclax (Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years.

  * Adults < 60 years are eligible if deemed unfit for intensive induction by their treating physician (or choose to receive a non-intensive regimen due to patient's preference)
* Diagnosis of treatment-naive AML (excluding acute promyelocytic leukemia treated with hydroxyurea) or high grade MDS defined as >10% marrow blasts or R-IPSS of intermediate 2 risk or higher with > 10% bone marrow blasts, and 1 or more of the following:

  * Circulating blasts in peripheral blood
  * Rapidly declining blood counts over the past 8 weeks, as determined by treating investigator
  * Transfusion dependence
  * Adverse cytogenetic changes or molecular mutations with high risk of rapid progression to AML, as determined by treating investigator
  * Significant B-symptoms attributed to MDS (weight loss, fatigue, unexplained fever, night sweats)
  * Evidence of clonal evolution with emergence of new cytogenetic changes or new mutations compared to previous bone marrow biopsy.
* White blood cell count < 25 K/uL. Cytoreduction with hydroxyurea is allowed prior to enrollment to obtain white blood cell count < 25 K/uL.
* Subjects of childbearing potential (SOCBP) must have a negative pregnancy test and agree to use of an adequate method of contraception to avoid pregnancy throughout the study and for at least 4 months after the last dose of study drug. Prior to study enrollment, subjects of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. Subjects with partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 4 months following the last dose of study drug.

Exclusion Criteria:

* Participants with acute promyelocytic leukemia (APML, APL, AML-M3)
* Patient with active central nervous system leukemia
* Karnofsky performance status < 50 at screening

  * Karnofsky performance status of 40-50 is allowed to proceed on study if the patient had a performance status of 50-100 at screening and the decline to 40 is deemed definitely related to disease (AML/MDS).
* Patients with AML with molecular mutations with FDA approved targeted therapies in the first line setting.

  * This includes FLT3 ITD/TKD + AML, IDH1+ AML. (Note: IDH2+ AML has targeted therapy approved in relapsed setting only; FDA approval for first line setting is pending and will be excluded once approval is obtained).
* Subjects with familial AML/MDS syndromes and those with inherited DNA repair syndromes like Fanconi Anemia
* Concurrent illness that in the opinion of the Investigator would pose an undue risk to the subject participating in this clinical study.
* Severe kidney impairment CrCL < 10 mL/min (per Cockcroft Gault equation) or dialysis-depended renal failure
* Class III-IV NYHA heart failure
* Child-Pugh class C liver cirrhosis
* Known seropositivity or active viral infection with human immunodeficiency virus (HIV), hepatis B virus (HBV), or hepatitis C virus (HCV) unless fully treated and negative by PCR. Patients who are seropositive because of HBV vaccine are eligible.
* Subjects with uncontrolled life-threatening infections

  * Subjects with fever (temperature > 38.3 C) thought to be related to AML/MDS are eligible
* History of allergic reaction to hypomethylating agents (decitabine, azacitidine), venetoclax, cladribine, or cytarabine.
* Active solid tumor malignancy requiring treatment within previous 2 years.

  * Patients with prior history of malignancy who completed treatment > 2 years prior to baseline are eligible to enroll if there is currently no evidence of disease and all toxicities of prior treatments are resolved.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Rate of complete remission | 18 months
  Compare the rate of complete remission (per 2017 European LeukemiaNet criteria for AML response assessment) in patients treated with cladribine/cytarabine alternating with decitabine to that for patients treated with decitabine or azacitidine and venetoclax

SECONDARY OUTCOMES:
Time to complete remission | 18 months
  Compare time to complete remission (per 2017 European LeukemiaNet criteria for AML response assessment) in patients treated with cladribine/cytarabine alternating with decitabine to that for patients treated with decitabine or azacitidine and venetoclax
Time to minimal residual disease (MRD) negativity | 18 months
  Compare time to MRD negativity (as measured by multicolor flow cytometry per current NCCN guidelines) in patients treated with cladribine/cytarabine alternating with decitabine to that for patients treated with decitabine or azacitidine and venetoclax
Overall survival | 30 months
  Compare overall survival (defined as the time from date of randomization until date of death) in patients treated with cladribine/cytarabine alternating with decitabine to that for patients treated with decitabine or azacitidine and venetoclax
Overall response rate | 18 months
  Compare overall response rate (defined as the number of patients who achieve either complete or partial remission per 2017 European LeukemiaNet criteria for AML response assessment) in patients treated with cladribine/cytarabine alternating with decitabine to that for patients treated with decitabine or azacitidine and venetoclax
Time to overall response | 18 months
  Compare time to overall response in patients treated with cladribine/cytarabine alternating with decitabine to that for patients treated with decitabine or azacitidine and venetoclax. Time to overall response is defined as the time interval from the date of treatment initiation to achievement of overall response.
Rate of MRD negativity | 18 months
  Compare rate of MRD negativity (as measured by multicolor flow cytometry per current NCCN guidelines) in patients treated with cladribine/cytarabine alternating with decitabine to that for patients treated with decitabine or azacitidine and venetoclax
Event-free survival | 30 months
  Compare event-free survival in patients treated with cladribine/cytarabine alternating with decitabine to that for patients treated with decitabine or azacitidine and venetoclax. Event-free survival is defined as the time from the date of randomization to induction treatment failure, relapse in those with a complete remission after induction, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crispen, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States